## **Statistical Analysis Plan Amendment 1**

**Study ID:** 212884

**Official Title of Study:** A phase IV, randomized, observer-blind, placebo-controlled, multi-center study to assess the prophylactic efficacy against Herpes Zoster, immunogenicity and safety of Shingrix when administered intramuscularly on a 2-dose schedule in Chinese adults aged 50 years and older

NCT number: NCT04869982

**Date of Document:** 10 May 2023

| Statistical Allalysis Flatt Afficiation | |
|---|---|
| , | Statistical Analysis Plan |
| Title: | A phase IV, randomized, observer-blind, placebo-<br>controlled, multi-center study to assess the<br>prophylactic efficacy against Herpes Zoster,<br>immunogenicity and safety of <i>Shingrix</i> when<br>administered intramuscularly on a 2-dose schedule in<br>Chinese adults aged 50 years and older |
| eTrack study number and<br>Abbreviated Title | 212884 (ZOSTER-076) |
| Scope: | All data pertaining to the above study. |
| Date of Statistical Analysis<br>Plan | Final: 08 February 2021 |
| 1 1411 | Amendment 1 Final: 10 May 2023 |
| APP 9000058193 Statistical Analysis Plan Template V5 (Effective date: 1July2020) | |

## 212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

## **TABLE OF CONTENTS**

| DOCUMENT HISTORY | | | | | PAGE |
|---|---|---|---|---|---|
| 2. OBJECTIVES/ENDPOINTS 8 3. STUDY DESIGN 10 4. ANALYSIS SETS 12 4.1. Definition 12 4.1.1. Enrolled Set 12 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3.1. Excluded subjects 14 4.2.3.1. Excluded subjects 14 4.2.4.2. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4.1. Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 18 5.4.1. Analysis of exposure planned in the protocol 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective <td>LIS</td> <td>T OF A</td> <td>ABBREVIA</td> <td>ATIONS</td> <td>6</td> | LIS | T OF A | ABBREVIA | ATIONS | 6 |
| 2. OBJECTIVES/ENDPOINTS 8 3. STUDY DESIGN 10 4. ANALYSIS SETS 12 4.1. Definition 12 4.1.1. Enrolled Set 12 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3.1. Excluded subjects 14 4.2.3.1. Excluded subjects 14 4.2.4.2. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4.1. Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 18 5.4.1. Analysis of exposure planned in the protocol 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective <td>1.</td> <td>DOCI</td> <td>JMENT H</td> <td>IISTORY</td> <td>7</td> | 1. | DOCI | JMENT H | IISTORY | 7 |
| 3. STUDY DESIGN 10 4. ANALYSIS SETS 12 4.1. Definition 12 4.1.1. Enrolled Set 12 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Exposed Set (ES) 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from Exposed Set (ES) 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4. Elimination from Unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.4.2. Additional considerations 17 5.4.2. Additional considerations 18 5.5.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity | | | | | |
| 4. ANALYSIS SETS 12 4.1. Definition 12 4.1.1. Enrolled Set 12 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Eprosed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.3. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective 18 5.5.1. Analysis of immunogenicity planned in the protoco | 2. | OBJE | CTIVES/I | ENDPOINTS | 8 |
| 4.1.1 Enrolled Set 12 4.1.2 Exposed Set 12 4.1.3 Modified Exposed Set 12 4.1.4 Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1 Elimination from Errolled Set 13 4.2.2 Elimination from Exposed Set (ES) 13 4.2.3 Ilimination from Per-prolocol analysis Set (PPS) 14 4.2.3.1 Excluded subjects 14 4.2.4.1 Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2 Subjects Disposition 17 5.3 Demography 17 5.3.1 Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2 Additional considerations 17 5.4 Exposure 18 5.4.1 Analysis of exposure planned in the protocol 18 5.5.1.1 Analysis of efficacy planned in the protocol 18 <td>3.</td> <td>STUE</td> <td>Y DESIG</td> <td>N</td> <td>10</td> | 3. | STUE | Y DESIG | N | 10 |
| 4.1.1 Enrolled Set 12 4.1.2 Exposed Set 12 4.1.3 Modified Exposed Set 12 4.1.4 Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1 Elimination from Errolled Set 13 4.2.2 Elimination from Exposed Set (ES) 13 4.2.3 Ilimination from Per-prolocol analysis Set (PPS) 14 4.2.3.1 Excluded subjects 14 4.2.4.1 Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2 Subjects Disposition 17 5.3 Demography 17 5.3.1 Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2 Additional considerations 17 5.4 Exposure 18 5.4.1 Analysis of exposure planned in the protocol 18 5.5.1.1 Analysis of efficacy planned in the protocol 18 <td>4.</td> <td>ANAL</td> <td>YSIS SE</td> <td>TS</td> <td>12</td> | 4. | ANAL | YSIS SE | TS | 12 |
| 4.1.1. Enrolled Set 12 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Errolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3. Additional considerations 17 5.4. Exposure 18 5.4. Analysis of exposure planned in the protocol 18 5.5. Efficacy/Effectiveness 18 5.5. Analysis of efficacy planned in the protocol 18 5.5. A | | | | | |
| 4.1.2. Exposed Set 12 4.1.3. Modified Exposed Set 12 4.1.4. Per Protocol Set 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.3.1. Excluded subjects 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective 18 5.5.1. <td></td> <td></td> <td></td> <td></td> <td></td> | | | | | |
| 4.1.3. Modified Exposed Set. 12 4.1.4. Per Protocol Set. 13 4.2. Criteria for eliminating data from Analysis Sets. 13 4.2.1. Elimination from Exposed Set (ES) 13 4.2.2. Elimination from modified Exposed Set (mES). 14 4.2.3. Elimination from modified Exposed Set (mES). 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4.1. Excluded subjects. 15 4.2.5. Elimination from unsolicited and solicited safety set. 16 5. STATISTICAL ANALYSES. 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol. 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5.1.1. Primary Objective 18 5.5.1. | | | | | |
| 4.1.4. Per Protocol Set. 13 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set. 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Excluded subjects 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4. Elimination from unsolicited subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5.1.1 Primary Objective 18 5.5.1.2 Secondary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 5.6.1. Analysis of immunogenicity planned in the protocol 20 5.6.2. Additional considerations 20 <td></td> <td></td> <td></td> <td></td> <td></td> | | | | | |
| 4.2. Criteria for eliminating data from Analysis Sets 13 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.3.1. Excluded subjects 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5. Efficacy/Effectiveness 18 5.5.1.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6.1. Analysis of immunogenicity planned in the protocol 20 5.6.2. Additional considerations 20 5.7. Analysis of safety and reactogenicity planned in the protocol 20 5.6.2. Additional considerations 20 | | | | | |
| 4.2.1. Elimination from Enrolled Set 13 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.3. Excluded subjects 14 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4.1. Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5.1. Primary Objective 18 5.5.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 </td <td></td> <td>12</td> <td></td> <td></td> <td></td> | | 12 | | | |
| 4.2.2. Elimination from Exposed Set (ES) 13 4.2.3. Elimination from modified Exposed Set (mES) 14 4.2.4. Elimination from Per-protocol 15 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.5.2. Additional considerations 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 5.6.2. Additional considerations 20 5.6.1. Analysis of immunogenicity planned in the protocol 20 5.6.2. Additional considerations 20 5.7.1. Analysis of safety and reactogenicity 21 5.7.2. Additional | | 4.2. | | | |
| 4.2.3. Elimination from modified Exposed Set (mES) | | | | | |
| 4.2.3.1. Excluded subjects | | | | | |
| 4.2.4. Elimination from Per-protocol analysis Set (PPS) 15 4.2.4.1. Excluded subjects 15 4.2.5. Elimination from unsolicited and solicited safety set 16 5.5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5. Efficacy/Effectiveness 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective 18 5.5.1.2. Secondary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 5.6.1. Analysis of immunogenicity 20 5.6.2. Additional considerations 20 5.7. Analysis of safety and reactogenicity 21 5.7.1. Analysis of safety and reactogenicity planned in the protocol 21 5.7.2. Additional considerations 22 5.7.2. Additional considerations 22 6. Analysis of safety and reactogenicity planned in the protocol 21 5.7.2. Additional considerations 22 6. Analysis of safety and reactogenicity planned in the protocol 22 5.6.2. Additional considerations 22 6. Analysis of safety and reactogenicity planned in the protocol 22 5.7.2. Additional considerations 22 6. Analysis of safety and reactogenicity planned in the protocol 22 5.7.2. Additional considerations 22 6. Analysis of safety and reactogenicity planned in the protocol 22 5.7.2. Additional 22 5.7.2. Additional 22 5.7.2. Additional 22 5.7.2. Additional 22 5 | | | 4.2.3. | | |
| 4.2.4.1. Excluded subjects | | | | | |
| 4.2.5. Elimination from unsolicited and solicited safety set 16 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1. Primary Objective 18 5.5.1. Primary Objective 18 5.5.1. Additional considerations 19 5.6. Immunogenicity 20 5.6.1. Analysis of immunogenicity planned in the protocol 20 5.6.2. Additional considerations 20 5.7.1. Analysis of safety and reactogenicity 21 5.7.1. Analysis of safety and reactogenicity planned in the protocol 21 5.7.2. | | | 4.2.4. | Elimination from Per-protocol analysis Set (PPS) | 15 |
| 5. STATISTICAL ANALYSES 16 5.1. General Considerations 16 5.2. Subjects Disposition 17 5.3. Demography 17 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol 17 5.3.2. Additional considerations 17 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5. Efficacy/Effectiveness 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 5.6.2. Additional considerations 20 5.7.1. Analysis of immunogenicity planned in the protocol 20 5.7.1. Analysis of safety and reactogenicity planned in the protocol 21 5.7.2. Additional considerations 22 6. ANALYSIS INTERPRETATION 23 | | | | | |
| 5.1.General Considerations165.2.Subjects Disposition175.3.Demography175.3.1.Analysis of demographics/baseline characteristics planned in the protocol175.3.2.Additional considerations175.4.Exposure185.4.1.Analysis of exposure planned in the protocol185.4.2.Additional considerations185.5.5.Efficacy/Effectiveness185.5.1.Analysis of efficacy planned in the protocol185.5.1.1.Primary Objective185.5.2.Additional considerations195.6.Immunogenicity205.6.1.Analysis of immunogenicity planned in the protocol205.6.2.Additional considerations205.7.Analysis of safety and reactogenicity215.7.1.Analysis of safety and reactogenicity planned in the protocol215.7.2.Additional considerations226.ANALYSIS INTERPRETATION23 | | | 4.2.5. | Elimination from unsolicited and solicited safety set | 16 |
| 5.2.Subjects Disposition.175.3.Demography.175.3.1.Analysis of demographics/baseline characteristics planned in the protocol175.3.2.Additional considerations175.4.Exposure185.4.1.Analysis of exposure planned in the protocol185.4.2.Additional considerations185.5.Efficacy/Effectiveness185.5.1.Analysis of efficacy planned in the protocol185.5.1.1.Primary Objective185.5.2.Additional considerations195.6.Immunogenicity205.6.1.Analysis of immunogenicity planned in the protocol205.6.2.Additional considerations205.7.1.Analysis of safety and reactogenicity planned in the protocol215.7.1.Analysis of safety and reactogenicity planned in the protocol215.7.2.Additional considerations226.ANALYSIS INTERPRETATION23 | 5. | | | | |
| 5.3. Demography | | _ | | | |
| 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol | | | | | |
| in the protocol | | 5.3. | | | |
| 5.3.2. Additional considerations | | | 5.3.1. | | |
| 5.4. Exposure 18 5.4.1. Analysis of exposure planned in the protocol 18 5.4.2. Additional considerations 18 5.5. Efficacy/Effectiveness 18 5.5.1. Analysis of efficacy planned in the protocol 18 5.5.1.1. Primary Objective 18 5.5.2. Additional considerations 19 5.6. Immunogenicity 20 5.6.1. Analysis of immunogenicity planned in the protocol 20 5.6.2. Additional considerations 20 5.7.1. Analysis of safety and reactogenicity 21 5.7.1. Analysis of safety and reactogenicity planned in the protocol 21 5.7.2. Additional considerations 22 6. ANALYSIS INTERPRETATION 23 | | | 500 | | |
| 5.4.1. Analysis of exposure planned in the protocol | | | | | |
| 5.4.2. Additional considerations | | 5.4. | • | | |
| 5.5. Efficacy/Effectiveness | | | | | |
| 5.5.1. Analysis of efficacy planned in the protocol | | | | | |
| 5.5.1.1 Primary Objective | | 5.5. | Efficacy | //Effectiveness | 18 |
| 5.5.1.2. Secondary Objective | | | 5.5.1. | | |
| 5.5.2. Additional considerations | | | | 5.5.1.1. Primary Objective | 18 |
| 5.6.Immunogenicity205.6.1.Analysis of immunogenicity planned in the protocol205.6.2.Additional considerations205.7.Analysis of safety and reactogenicity215.7.1.Analysis of safety and reactogenicity planned in the protocol215.7.2.Additional considerations226.ANALYSIS INTERPRETATION23 | | | | 5.5.1.2. Secondary Objective | 18 |
| 5.6.Immunogenicity205.6.1.Analysis of immunogenicity planned in the protocol205.6.2.Additional considerations205.7.Analysis of safety and reactogenicity215.7.1.Analysis of safety and reactogenicity planned in the protocol215.7.2.Additional considerations226.ANALYSIS INTERPRETATION23 | | | 5.5.2. | Additional considerations | 19 |
| 5.6.1. Analysis of immunogenicity planned in the protocol | | 5.6. | Immund | ogenicity | 20 |
| 5.6.2. Additional considerations | | | | | |
| 5.7. Analysis of safety and reactogenicity | | | | | |
| 5.7.1. Analysis of safety and reactogenicity planned in the protocol | | 5.7 | | | |
| protocol | | 0.7. | • | | |
| 5.7.2. Additional considerations | | | | | 21 |
| 6. ANALYSIS INTERPRETATION | | | 5.7.2. | | |
| | | | | | · — <del>-</del> |
| 7 INTEDIM ANALYSES 24 | 6. | ANAL | YSIS INT | ERPRETATION | 23 |
| | 7 | INITE | DINA ANIAI | VSES | 24 |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1 Sequence of analyses......24 7.1. 7.2. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS.......25 NON-STANDARD DATA DERIVATION RULES AND STATISTICAL 9.1. Demography ......25 9.1.1. 9.2. HZ incidence......26 9.2.1. 9.2.3. 10.1. Business rules for standard data derivations and statistical methods.......37 10.1.1. Handling of missing data......37 10.1.2. 10.1.2.3.1. Studies with electronic diaries.................38 10.1.2.3.2. Studies with paper diaries.......................38 10.1.2.4. 10.1.3. 10.1.3.1. Age at first dose in years ......40 10.1.3.2. Temperature......40 Onset day......40 10.1.3.3. Duration of events ......40 10.1.3.4. 10.1.3.5. Counting rules for combining solicited and unsolicited adverse events ......40 Counting rules for occurrences of solicited 10.1.3.6. events.....41 10.1.4. 10.1.4.1. Percentages .......41 10.1.4.2. Demographic/baseline characteristics statistics .........41 10.1.5. Statistical methodology......41 10.1.5.1. Exact confidence intervals around proportions .........41 TFL TOC......41 10.2.

11 REFERENCES 41

## 212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

## LIST OF TABLES

| | | PAGE |
|---------|---------------------------------------------------|------|
| Table 1 | Number of subjects required for enrolment | 11 |
| Table 2 | Intervals between study visits applicable for PPS | 13 |
| Table 3 | Intensity scales for solicited symptoms in adults | 28 |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

## LIST OF FIGURES

| | | PAGE |
|----------|-----------------------|------|
| Figure 1 | Study design overview | 10 |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

## List of abbreviations

AE Adverse event

AAC All Analyses Complete
CI Confidence Interval

CRF Case Report Form

CTRS Clinical Trial Registry Summary

EoS End of Study
ES Exposed Set

gE VZV glycoprotein E GM Geometric Mean

GSK GlaxoSmithKline Biologicals SA

HZ Herpes Zoster

HZAC HZ Ascertainment Committee

ICF Inform Consent Form ICS Intracellular staining

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

mES Modified Exposed Set

PBMC Peripheral Blood Mononuclear Cells

PCR Polymerase Chain Reaction

pIMD Potential Immune-Mediated Disease

PPS Per Protocol Set

RAPIDO DV Reporting & Analysis Plan Improving Design and Delivery of

Outputs Data Viewer

RR Relative Risk

RZV Recombinant Zoster Vaccine

SAE Serious adverse event SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomisation System

SD Standard Deviation

SDTM Study Data Tabulation Model

SR Study Report

TFL Tables Figures and Listings

TOC Table of Content
VE Vaccine Efficacy
YOA Years of Age

## 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 08 FEB 2021 | Initial Version | Amendment 2 Final: 23 NOV 2020 |
| 10 May 2023 | Amendment 1: Following are the changes from SAP from 08 FEB 2021:- Added RAPIDO DV Added analysis of deviation from protocoldefined age and visit interval on ES. Updated model of vaccine efficacy: added by agecat statement and removed agecat from model. Substituted kaplan meier curves by cumulative incidence curves. Calculation and derivation rule for some solicited adverse event grade 4 and duration has been added Related grade 1 and related grade 2 have been added to GSK and Chinese scale analyses. Substituted 'grade 3' by at 'least grade 3' in solicited local and solicited general summaries based on GSK scale. Also, added the categories that will be displayed for fever in solicited general summaries Update of grade 3 definition for redness and swelling based on Chinese scale Update of the Preferred Terms used to determine grade 4 for Redness and Swelling. Update in handling of missing data in section 10.1.2.3.2 Analysis for secondary safety endpoint related to 'SAE due to study participation and GSK concomitant medication/vaccination' has been added. Analysis of concomitant medication related to confirmed HZ episode has been added Covid-19 related analyses have been added Minor edits in text for clarification. Added site specific Covid-19 pandemic measure periods | Amendment 2 Final: 23 NOV 2020 |

## 2. OBJECTIVES/ENDPOINTS

Below are the study objectives and endpoints:-

| Objectives | Endpoints |
|---|---|
| P | rimary |
| To evaluate vaccine efficacy (VE) in the prevention of HZ compared to placebo in Chinese adults ≥ 50 YOA, as measured by the reduction in herpes zoster (HZ) risk. **Criterion:* The objective is met if the lower limit (LL) of the 2-sided 95% confidence interval (CI) of VE is above 25%. | Confirmed HZ cases in the modified Exposed Set (mES). |
| Se | condary |
| To evaluate VE in the prevention of HZ compared to placebo in subjects within each of the following age ranges: 50-69 years of age (YOA) and <sup>3</sup> 70 YOA, as measured by the reduction in HZ risk | Confirmed HZ cases within each of the following age ranges: 50-69 YOA and <sup>3</sup> 70 YOA in the mES. |
| To evaluate vaccine reactogenicity and safety | <ul> <li>Solicited local and general adverse events (AEs)</li> <li>Occurrence, intensity and resulting in medically attended visit of each solicited local AE within 7 days (Days 1 – 7) after each vaccination</li> <li>Occurrence, intensity and resulting in medically attended visit and relationship to</li> </ul> |
| | vaccination of each solicited general AE within 7 days (Days 1 – 7) after each vaccination. |
| | Unsolicited AEs |
| | Occurrence, intensity, resulting in a medically-attended visit, and relationship to vaccination of unsolicited AEs (including cellulitis) within 30 days (Days 1 – 30) post-vaccination period, according to the Medical Dictionary for Regulatory Activities (MedDRA) classification. |
| | Serious Adverse Events (SAEs) Occurrence and relationship to vaccination of SAEs from Day 1 up to 30 days post last vaccination. |

## 3. STUDY DESIGN

Figure 1 Study design overview



; N= number of subjects planned to be enrolled; Vacc= Vaccination

RZV= Recombinant Zoster Vaccine

‡ All subjects will be followed-up until last enrolled subject has completed 1 year of follow-up post last vaccination. In case criteria for vaccine efficacy analyses are not met during this period, the follow-up will be extended.

- **Experimental design**: Phase IV, randomized, observer-blind, placebo-controlled, multi-centric, single-country study with 2 parallel groups.
- **Duration of the study:** The duration of the study will vary for each subject. The duration of the study will be up to the study conclusion contact that occurs within 30 days of the projected study conclusion date of the last enrolled subject, that is, 14 months (approximately 430 days) from the enrolment date. Therefore, subjects enrolled early in the trial will be followed for longer duration than the subjects who enrol later in the trial. In case criteria for VE analyses are not met during this period, the follow-up will be extended.

The study conclusion visit/ contact for subjects with an ongoing episode of HZ at the time of last subject last contact will occur at Visit HZ-5 (Day HZ-29).

- Epoch 001 (Vaccination phase): Starting at Visit 1 (Day 1) until Visit 3 (Month 3) at one month post last vaccination.
- Epoch 002 (Follow-up phase): Starting with the first monthly contact after
   Visit 3 (Month 3) and ending at the monthly contact that occurs within 30 days
   of the projected study conclusion date of the last enrolled subject, that is, 14
   months (approximately 430 days) from the enrolment date of the last enrolled
   subject.
- **Primary completion Date (PCD):** The primary completion date will be when the last subject completes his/her study conclusion contact (within 30 days of the projected study conclusion date of the last enrolled subject, that is, 14 months (approximately 430 days) from the enrolment date. In case criteria for VE analyses are not met during this period, the follow-up will be extended.

212884 (ZOSTER-076)

Statistical Analysis Plan Amendment 1

- End of Study (EoS): 1) After all the subjects complete their study conclusion contact, occurring within 30 days of the projected study conclusion date of the last enrolled subject, that is, 14 months (approximately 430 days) from the enrolment date of the last subject; In case criteria for VE analyses are not met during this period, the follow-up will be extended and 2) the release of all polymerase chain reaction (PCR) test results for the HZ rash lesion samples. Refer to section 7.1 for more detail.
- Control: placebo controlled
- **Vaccination schedule**: 0 and 2 months
- Treatment allocation: Eligible subjects will be randomized (1:1) to RZV group or Placebo group. The randomization algorithm will use a stratification procedure accounting for age (50-69 YOA and≥ 70 YOA).
- Sampling schedule:
  - CCI
  - Clinical specimens of HZ lesions will be collected from all subjects who are clinically diagnosed with a suspected case of HZ (Section 8.3.2 of the protocol).
  - A urine specimen will be collected from all female subjects of child-bearing potential (see glossary of terms in the protocol definition of woman of child bearing potential) at Visit 1 (Day 1) and Visit 2 (Month 2).
- Study group and treatment number allocation: The target will be to enrol approximately 6138 eligible subjects who will be randomly assigned to 2 study groups in a (1:1) ratio (approximately 3069 subjects in each group).

The enrolment will be performed to ensure distribution of the population across the 2 age strata (50-69 YOA and  $\geq$ 70 YOA). Approximately 75-80% and 20-25% subject should be enrolled in 50-69 YOA and  $\geq$ 70 YOA, respectively. The expected distribution of subjects within these 2 age strata is as shown in Table 1.

To ensure that the collection of date of birth will not jeopardize the privacy of Personally Identifiable Information (PII), only year of birth (YYYY) will be collected.

Table 1 Number of subjects required for enrolment

| | Age Stratum | Vaccine | Targeted number (%) of subjects |
|---|-------------|--------------------|---------------------------------|
| ſ | 50-69 YOA | RZV 4004 4040 (75) | |
| | 50-69 YOA | Placebo | 4604-4910 (75-80%) |
| | ≥ 70 YOA | RZV | 1000 1524 (00 050) |
| | ≥ 10 YUA | Placebo | 1228-1534 (20-25%) |

Allocation of the subject to a study group at the investigator site will be performed using a randomization system on internet (SBIR). Within each age stratum, the randomization algorithm will use a minimization procedure accounting for center, gender, age (50-59, 60-69, 70-79 and ≥80 YOA) and a combined minimization factor to reflect the presence of any of the following conditions: type 2 diabetes mellitus, asthma, chronic obstructive pulmonary disease, chronic kidney disease and depression. Minimization factors will have equal weight in the minimization algorithm.

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

| • | Allocation of subjects to assay subsets - CCI |
|-----|-----------------------------------------------|
| CCI | |

## 4. ANALYSIS SETS

## 4.1. Definition

#### 4.1.1. Enrolled Set

The enrolled set will include all eligible subjects who have signed an informed consent and were randomized or undergone an invasive procedure.

## 4.1.2. Exposed Set

Exposed Set (ES) will include all subjects who receive at least 1 dose of the study treatment. The allocation in a group is done in function of the administered treatment.

The ES for the analysis of solicited AEs will include all participants who received at least 1 dose of the study treatment and who have documented solicited AEs (i.e. diary card for solicited AEs completed and returned).

The ES for the analysis of any other AEs other than solicited AEs will include all participants who received at least 1 dose of the study treatment.



## 4.1.3. Modified Exposed Set

The modified Exposed Set (mES) excludes subjects from the ES who were not administered 2 doses of the study treatment per protocol, or who developed a confirmed case of HZ prior to 30 days after the second vaccination (Refer to section 4.2.3 for more detail on the criteria).

#### 4.1.4. Per Protocol Set

All subjects who received at least 1 dose of the study treatment to which they are randomised and have post-vaccination data minus subjects with protocol deviations that lead to exclusion. The Per Protocol Set (PPS) (in vaccinated subjects) will include all evaluable vaccinated subjects:

- CCI
- who have received 2 doses of study vaccine;
- for whom the study vaccine has been administered as per protocol;
- who have not received medication/vaccine forbidden in the protocol (refer to Section 4.2.4 for details on the criteria);
- who meet all eligibility criteria (refer to Sections 6.1 and 6.2 of the protocol);
- who comply with the procedures and intervals defined in the protocol;
- who do not meet any of the criteria for elimination during the study (refer to Section 4.2.4 for details on the criteria);
- for whom data concerning immunogenicity endpoint measures are available.

The intervals allowed for the inclusion in the PPS is the 'allowed interval per protocol' as defined in following table:

Table 2 Intervals between study visits applicable for PPS

| Interval | Optimal length of interval | Allowed interval per protocol |
|-----------------|----------------------------|-------------------------------|
| Visit 1→Visit 2 | 60 days (2 months) | 49 days - 83 days |
| Visit 2→Visit 3 | 30 days (1 month) | 28 days - 48 days |

## 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

#### 4.2.1. Elimination from Enrolled Set

Code 800 (fraudulent data), 900 (invalid ICF) and 1010 (treatment number not allocated) will be used for identifying subjects eliminated from Enrolled Set.

## 4.2.2. Elimination from Exposed Set (ES)

Code 1030 (Study treatment not administered at all), 800 (fraudulent data), 900 (invalid ICF) and 1010 (treatment number not allocated) will be used for identifying subjects eliminated from ES.

Statistical Analysis Plan Amendment 1

## 4.2.3. Elimination from modified Exposed Set (mES)

Code 1030 (Study treatment not administered at all), 800 (fraudulent data), 900 (invalid ICF), 1010 (treatment number not allocated), 1070 (treatment not administered according to protocol), 2500 (Subject who didn't receive two doses) and 3500 (Subject having confirmed HZ episode prior to 30 days after the dose 2) will be used for identifying subjects eliminated from mES.

Please note that impact of COVID-19 on the modified Exposed Set for vaccine efficacy analysis will be determined on a case-by-case basis.

## 4.2.3.1. Excluded subjects

A subject will be excluded from the mES analysis under the following conditions. Please note that impact of COVID 19 on the mES will be determined on a case-by-case basis.

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable |
|---|---|---|
| 800 | Fraudulent data | All |
| 900 | Invalid ICF | Visit 1 |
| 1010 | Treatment number not allocated | Visit 1 |
| 1030 | Study vaccine not administered at all | Visit 1 |
| 1070** | Vaccination not according to protocol: | Visit 1, Visit 2 |
| | <ul> <li>Subjects got vaccinated with the correct vaccine but containing a lower volume</li> <li>Administration not according to protocol for reason specified by investigator other than route, side and site.</li> <li>Site and route of vaccination is wrong or unknown</li> <li>Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number)</li> </ul> | |
| 2500 | Subjects who didn't receive two doses | Visit 2 |
| 3500 | Subjects having confirmed HZ episode prior to 30 days after the dose 2 | Visit 1 to Visit 3 |

<sup>\*\*</sup> Attribution of these elimination codes will be evaluated on case-by-case basis and requires CRDL confirmation

## 4.2.4. Elimination from Per-protocol analysis Set (PPS)

## 4.2.4.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions. Please note that impact of COVID 19 on the per protocol set will be determined on a case-by-case basis.

| Code | Condition under which the code is used | Visit (timepoints) where the code is applicable |
|---|---|---|
| 800 | Fraudulent data | All |
| 900 | Invalid ICF | Visit 1 |
| 1010 | Treatment number not allocated | Visit 1 |
| 1030 | Study vaccine not administered at all | Visit 1 |
| 1040* | Administration of concomitant vaccine(s) | - 30 days to Visit 1 |
| | forbidden in the protocol | through Visit 3 |
| | Any concomitant vaccination not foreseen by the | _ |
| | study protocol administered in the period starting | |
| | 30 days before the first dose of the study vaccine | |
| | and ending at Visit 3 (Day -30 to Month 3) | |
| 1050 | Randomisation failure | A11 |
| 1060 | Randomisation code was broken | Visit 1 to Visit 3 |
| 1070** | Vaccination not according to protocol: | Visit 1, Visit 2 |
| | Subjects got vaccinated with the correct | |
| | vaccine but containing a lower volume | |
| | Administration not according to protocol for | |
| | reason specified by investigator other than | |
| | route, side and site. | |
| | Site and route of vaccination is wrong or | |
| | unknown | |
| | Wrong replacement or study vaccine | |
| | administered (not compatible with the vaccine | |
| | regimen associated to the treatment number) | |
| 1080 | Vaccine temperature deviation | Visit 1, Visit 2 |
| 1090 | Expired vaccine administered | Visit 1, Visit 2 |
| 2010 | Protocol violation (inclusion/exclusion criteria) | Visit 1 |
| 2040* | Administration of any medication forbidden by the | Visit 1 to Visit 3 |
| | protocol (refer to Section 7.5.2 of the protocol) | |
| | administered in the period from the first dose of | |
| | study vaccine and ending at Visit 3 (Day 1 to | |
| | Month 3) | |

Statistical Analysis Plan Amendment 1

| Code | Condition under which the code is used | Visit (timepoints) where the code is |
|---|---|---|
| | | applicable |
| 2050* | Underlying medical condition forbidden by the protocol | Visit 1 to Visit 3 |
| | Any intercurrent medical condition (IMC) (refer to | |
| | section 7.6 of the protocol) which can affect the | |
| | immune response to the study vaccine and ending at Visit 3 (Day 1 to Month 3) | |
| 2060* | Concomitant infection related to the vaccine which may influence immune response | Visit 1 to Visit 3 |
| 2070* | Concomitant infection not related to the vaccine which may influence immune response | Visit 1 to Visit 3 |
| 2080 | Subjects did not comply with vaccination schedule $DOSE\ 1 - DOSE\ 2 = 49-83\ days$ | Visit 2 |
| 2090 | Subjects did not comply with blood sample schedule DOSE2 - blood sample (BS)2 = 28-48 days | Visit 3 |
| 2100 | Serological results not available post-vaccination | Visit 3 |
| 2120 | Obvious incoherence or abnormality or error in data | Visit 3 |
| 2500 | Subjects who didn't receive two doses | Visit 2 |
| 3500 | Subjects having confirmed HZ episode prior to 30 days after the dose 2 | Visit 1 to Visit 3 |
| 2130 | CCI | |

<sup>\*</sup>Attribution of these elimination codes to subject need CRDL review of individual listing

# CCI

## 4.2.5. Elimination from unsolicited and solicited safety set

Unsolicited and solicited safety set is not applicable for the study.

## 5. STATISTICAL ANALYSES

The standard data derivation rules and stat methods are described in section 10.1 while the study specific data derivation rules and stat methods are described in section 9 of the SAP.

Analysis on Covid-19 cases has been added in the analysis of safety section of the SAP.

## 5.1. General Considerations

Note: Subject-level data will be available interactively via RAPIDO DV after AAC.

<sup>\*\*</sup> Attribution of these elimination codes will be evaluated on case-by-case basis and requires CRDL confirmation

## 5.2. Subjects Disposition

Number of enrolled and vaccinated (at least 1 vaccination) subjects, included in each group or in total for a given age category or for all age categories will be described.

## 5.3. Demography

## 5.3.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic and other baseline characteristics will be described by assigned group and for the total for ES and mES and the CCI.

Demographic characteristics (age at first study vaccination in years, gender, race and ethnicity) will be summarized overall and by study groups using descriptive statistics:

- Frequency tables will be generated for categorical variables such as center.
- Mean, standard deviation, median, minimum and maximum will be provided for continuous data such as age.

Cohort description and withdrawal status will be summarized by group and overall. All important protocol deviations leading to elimination will be presented.

All the above analyses will be performed by age strata (50-69 YOA and  $\geq$  70 YOA) on ES and mES.

### 5.3.2. Additional considerations

Following additional tables will also be generated:

- Number of subjects by centers will be presented on ES.
- Deviation from protocol-defined age and visit interval on ES.
- The following table will be generated for web disclosure:
  - Percentage of enrolled subjects by age categories (18-64, 65-84, ≥85) YOA will be tabulated by group.
- Summary of important protocol deviations leading to elimination from any analysis will be presented for the Enrolled Set overall and by age strata.
- The number of subjects enrolled into the study as well as the number of subjects excluded from *mES and* PPS analyses will be presented through 3 consort tables, overall and by age strata only for Consort table 1 and 2:
  - Consort table 1 Showing the subjects disposition from Enrolled Set to ES
  - Consort table 2 Showing the subjects disposition from ES to mES
  - Consort table 3 Showing the subjects disposition from ES to PPS

## 5.4. Exposure

## 5.4.1. Analysis of exposure planned in the protocol

None

#### 5.4.2. Additional considerations

The number of doses administered will be tabulated. The number of doses administered will be tabulated by age stratum.

## 5.5. Efficacy/Effectiveness

The primary analysis of efficacy will be based on the mES. A secondary analysis based on the ES will performed to complement the mES analysis.

## 5.5.1. Analysis of efficacy planned in the protocol

## 5.5.1.1. Primary Objective

The primary inferential analysis of efficacy on the mES will be based on the occurrence of the primary endpoint anytime from 30 days after the administration of the second dose of the study vaccine up to study end. All subjects from the mES will contribute to the comparison.

It will consider the exact inference on the relative risk (RR) adjusted for age strata conditionally to the total number of HZ cases observed and time at risk. This method computes an exact CI around the rate ratio (ratio of the event rates in the RZV group versus control group) and takes into account, the sum of the time at risk of the subjects within each group.

Incidence rate and VE with 95% CI will be calculated using Poisson method. The VE will be defined as 1 minus the RR. RR is defined as the ratio of the incidence rates of the RZV group over the placebo group [VE=  $(1 - RR) \times 100$ ]

The VE of RZV against HZ will be demonstrated if the LL of the two-sided 95% CI of VE is above 25%. All p-values reported will be related to the null hypothesis test VE = 0.

The calculation of the time at risk and other statistical method detail are provided in Section 9.2.1.

## 5.5.1.2. Secondary Objective

The number of confirmed HZ cases, follow-up days, associated rate, VE with 95% CI will be presented by each age category, descriptively, as for the primary endpoint.

## 5.5.2. Additional considerations

Following descriptive table and figure will be generated by study groups on mES and ES:

- For each study group, the number of subjects at risk, person-year, number and incidence of confirmed HZ will be tabulated overall.
- Forest plot for vaccine efficacy against HZ by age strata and overall during the entire study period
- Cumulative incidence curve for HZ for each study group.
- Number and percentage of episodes of all confirmed HZ episodes during the entire study period.
- Number and percentage of confirmed HZ episodes out of all the suspected cases reported.
- Number and percentage of suspected cases for which at least one PCR sample was collected on ES only.
- Distribution of suspected HZ cases using the HZ classification tools (PCR testing & HZ Ascertainment Committee (HZAC))
- The vaccine efficacy will be assessed by Poisson method for primary objective and fitted via the PROC GENMOD procedure according to the following code

```
PROC GENMOD DATA=pois ve EXACTONLY;
BY AGECAT;
STRATA AGECAT:
CLASS AGECAT/PARAM=ref;
MODEL nb cases = group nb/DIST=poisson OFFSET = Log T LINK=log;
EXACT group nb/ESTIMATE OUTDIST=dist ALPHA=0.05;
ODS OUTPUT ExactParmEst=estimate ExactTests=ExactTest:
RUN;
Where,
nb case = number of cases
agecat = Age strata categories (50-69 and \geq=70 YOA)
group nb = Group information of the subject (treatment received by subject)
Log T = Log of the follow-up time
DATA VE;
SET ESTIMATE;
FORMAT VE best12. Il best12. ul best12.;
VE = (1 - exp (estimate)) * 100;
11 = (1 - \exp(UPPERCL)) * 100;
ul = (1 - exp(LOWERCL)) * 100;
RUN:
```

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1



## 5.6.2. Additional considerations

None

Statistical Analysis Plan Amendment 1

## 5.7. Analysis of safety and reactogenicity

## 5.7.1. Analysis of safety and reactogenicity planned in the protocol

The primary analysis of safety will be performed on the ES. All analyses will also be performed by age strata (50-69 YOA and  $\geq$ 70 YOA). Following analysis is planned to be performed:

The percentage of subjects with at least 1 local AE (solicited and unsolicited), with at least 1 general AE (solicited and unsolicited) and with any AE (solicited and unsolicited) during the solicited follow-up period will be tabulated with exact 95% CI after each vaccine dose and overall. The percentage of doses followed by at least 1 local AE (solicited and unsolicited), by at least 1 general AE (solicited and unsolicited) and by any AE will be tabulated, with exact 95% CI. The percentage of subjects with at least 1 local AE (solicited only), with at least one general AE (solicited only) and with any AE (solicited only) during the solicited 7-day follow-up period will be tabulated with exact 95% CI after each vaccine dose and overall.

The percentage of subjects reporting each solicited local and general AE during the solicited follow-up period will be tabulated with exact 95% CI. The percentage of doses followed by each individual solicited local and general AE will be tabulated, with exact 95% CI. Fever will be reported with any (>=38.0), >=38.0 - <=38.5, >38.5 - <=39.0 and >39.0 in GSK scale. In Chinese scale, it will be reported with any (>=37.3), 37.3 - <38.0, 38.0 - <38.5, 38.5 - <39.5 and >=39.5. The same tabulation will be performed for fever with causal relationship to the study vaccine.

In the table presented based on the GSK scale, for all other solicited AEs, the same table will have grade 1, grade 2 and at least grade 3 AEs and for any and at least grade 3 general AEs with relationship to the study vaccine. Related grade 1 and related grade 2 will also be displayed.

In the table presented based on the Chinese scale, for all other solicited AEs, the same table will have grade 1, grade 2, grade 3 and grade 4 applicable for table with Chinese intensity scale) AEs and for any, grade 3 and grade 4 general AEs with relationship to the study vaccine. Related grade 1 and related grade 2 will also be displayed.

The proportion of solicited AEs resulting in a medically attended visit will be tabulated.

The percentage of subjects with at least 1 report of unsolicited AE (including cellulitis) classified by MedDRA primary system organ class (SOC) and preferred terms (PT) will be reported within 30 days (Days 1-30) post each vaccination with exact 95% CI. The same tabulation will be performed for grade 3 unsolicited AEs, for unsolicited AEs with a relationship to vaccination, grade 3 unsolicited AEs with a relationship to vaccination.

Number and percentage of any, grade 3, related, grade 3 related and medically attended unsolicited AEs reported within 30 days (Days 1-30) post *any* vaccination according to MedDRA primary system organ class and preferred terms will be presented.

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

Number and percentage of SAEs from first vaccination up to 12 months post last vaccination will be presented with 95% CI. The same tabulation will also be done for the interval- starting from first vaccination up to 30 days post last vaccination.

Number and percentage of SAEs causally related to vaccination for the interval-starting from first vaccination up to 30 days post last vaccination and from first vaccination up to 12 months post last vaccination and from study start up to study end will be presented with 95% CI.

Number and percentage of subjects experiencing fatal SAEs, classified by MedDRA Primary System Organ Class and Preferred Term will be tabulated using date of onset of SAE for the time periods –from first vaccination up to 30 days post last vaccination and first vaccination up to 12 months post last will be presented with 95% CI.

Number and percentage of fatal SAEs causally related to vaccination for the intervalstarting from first vaccination up to 30 days post last vaccination and from first vaccination up to 12 months post last vaccination and from study start up to study end will be presented with 95% CI.

Number and percentage of pIMDs from first vaccination up to 12 months post last vaccination will be presented with 95% CI. The same tabulation will also be done for the interval – starting from first vaccination up to 30 days post last vaccination.

Number and percentage of pIMDs causally related to vaccination from first vaccination up to 12 months post last vaccination will be presented with 95% CI. The same tabulation will also be done for the interval – starting from first vaccination up to 30 days post last vaccination. Number and percentage of serious pIMDs causally related to vaccination from 12 months post last vaccination up to study end and will be presented with 95% CI.

The proportion of subjects with concomitant medication will be tabulated, within 30 days post each vaccination and overall only, with exact 95% CI.

Listing of fatal SAEs, SAEs, pIMDs and withdrawals (from the study or from vaccination) due to AEs, SAEs, solicited and unsolicited AEs will be generated.

Listing of pregnancy during the entire study period will be generated.

Listing for all the suspected HZ episodes will be generated.

## 5.7.2. Additional considerations

The table on solicited local and general AEs will be presented separately according to GSK grading and grading scale provided by Chinese authorities.

Duration of each solicited local and general AE during the solicited follow-up period will be presented. Total duration of each individual solicited local and general AE will be tabulated.

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

Duration of each grade 3 solicited local and general AE during the solicited follow-up period will be presented in the table by GSK grading. Duration of each grade 3 and above solicited local and general AE during the solicited follow-up period will be presented in the table by Chinese authority grading.

Listing of complication related to confirmed HZ episode will be presented.

Number and percentage of subjects experiencing fatal SAEs, classified by MedDRA Primary System Organ Class and Preferred Term will be tabulated using date of onset of SAE from study start up to study end will be presented with 95% CI for web disclosure.

The table for web disclosure related to *solicited adverse events* endpoint will be based on both GSK and Chinese intensity scale.

Summary of subjects with serious adverse events related to study participation and not by the study vaccines or to GlaxoSmithKline concomitant medication/vaccine during the entire study period based on ES.

Following listings of concomitant medications related to confirmed HZ episode will be presented based on Exposed Set:

- Pain rescue medication to control HZ pain
- Antiviral treatment for HZ
- Other therapy for HZ

Additional analyses/considerations due to COVID-19 pandemic on ES:

- Summary of COVID-19 Assessment.
- Incidence of COVID-19 as an AE and SAE. A standardized MedDRA Query (SMO) will be used to identify all COVID-19 cases reported as AEs.
- A column to identify COVID-19 AEs/SAEs will be added to listing of (S)AEs and solicited adverse events leading to study or treatment discontinuation from first vaccination up to study end.

## 6. ANALYSIS INTERPRETATION

The primary objective of VE in the prevention of HZ compared to placebo in Chinese adults≥ 50 YOA, as measured by the reduction in HZ risk is considered met if the LL of the 2-sided 95% CI of VE is above 25%.

For all secondary objectives, analyses will be descriptive with the aim to characterize the differences in reactogenicity, safety and immunogenicity between groups.

## 7. INTERIM ANALYSES

## 7.1. Sequence of analyses

The analysis of all primary and secondary endpoints will be performed when all data up to study conclusion are available. A clinical study report (CSR) will be written at this stage and individual listings will be included.

One final analysis is planned and will be triggered when the following will take place:

- When at least 27 confirmed cases of HZ have accrued in the primary cohort for efficacy (cut-off date for primary efficacy analysis); AND
- When all subjects have completed at least 12 months safety follow-up post last vaccination.

Data contributing to the analysis of the primary efficacy objective (confirmed HZ cases) will be collected until the cut-off date. After the cut-off date, case confirmation of any new suspected HZ will not be performed. Once the study reaches the cut-off date, the conclusion contact for a subject will be planned based on the status of the safety follow-up:

- Cut-off date reached before the completion of safety follow-up Continue the monthly safety follow-up after the cut-off date until all subjects have completed 12 months of follow-up post last dose.
- Cut-off date reached after the completion of safety follow-up Continue the monthly contacts after the completion of the 12 months safety follow-up period until at least 27 confirmed HZ cases have accrued (cut-off date).

When the trigger for primary efficacy analysis is reached, subjects with an ongoing HZ episode will be followed until Day HZ-29.

The conclusion contact of the last subject will be the study end.

If the data for exploratory endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These analyses will be documented in the annex study report.

| • | Disclosure Purpose (CTRS=public posting, SR=Study report, internal) |
|-------|---------------------------------------------------------------------|
| Final | Public disclosure, Study report |

## 7.2. Statistical considerations for interim analyses

No interim analysis will be performed.

Statistical Analysis Plan Amendment 1

# 8. CHANGES TO THE PROTOCOL DEFINED STATISTICAL ANALYSIS

Following is the change from protocol defined statistical analysis:-

- Fatal SAEs will not be tabulated using the date of death within the same time periods.
- CCI
- Grade 3 for redness/swelling will be defined as redness/swelling with diameter
   =100 mm in Chinese scale
- Preferred Terms to identify Grade 4 for swelling and redness have been added
- The analysis on at least 1 local AE (solicited and unsolicited; solicited only) with at least 1 general AE (solicited and unsolicited; solicited only) and with any AE (solicited and unsolicited; solicited only) during the solicited follow-up period with causal relationship with vaccine and AE rated as at least grade 3 according to GSK and Chinese scale will not be performed.

## 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1.

#### 9.1. Data derivation

## 9.1.1. Demography

For computation of age, following rule need to be considered:

- Age will be calculated as the number of years between the date of birth and the date of first vaccination.
- To ensure that the collection of date of birth will not jeopardise the privacy of Personal Identifiable Information (PII), only a partial date of birth (YYYY) will be collected. As the date and month will be missing, the date will be replaced by the June 30th of the year.

## 9.2. Statistical Method

#### 9.2.1. HZ incidence

- For the primary analysis of HZ incidence, first confirmed HZ episode will be considered.
- The HZ onset date is the earlier of the following two events: 1) the HZ rash start date; or 2) the date on which pain/itching or abnormal sensation at the site of a subsequent HZ rash is first noted.
- A suspected case of HZ can be confirmed by GSK in two ways:
  - **By PCR**: Rash lesion samples will be collected from subjects clinically diagnosed as having a suspected case of HZ. The samples will be transferred to GSK or a validated laboratory designated by GSK Biologicals and analyzed using standardized and validated procedures for laboratory diagnosis of HZ by PCR (see Section 12.2 of the protocol).
  - be referred to the HZAC. The HZAC will classify all referred cases as either "HZ" or "not HZ" or "not able to decide" (see Section 12.2 of the protocol). The HZAC classification will serve as the final case definition only when the case cannot be confirmed or excluded by PCR. Therefore, definitive PCR results, when available, will determine the final HZ case assignment. In such cases, the HZAC classification will not contribute to HZ case determination decision
- For a given subject and for HZ episode, missing or non-evaluable measurements will not to be imputed for the primary analysis. The missing endpoint and censoring are considered to occur independently, and the pattern being either Missing Completely At Random (MCAR) or Missing At Random (MAR) only.
- For HZ analysis, due to the algorithm used and taking into account both laboratory and HZAC results, no imputation and no sensitivity analysis for missing data will be performed.
- The "follow-up time at risk" for confirmed HZ is expressed in days and is computed according to the following rules:
  - The start date of the follow-up time (start) will be computed as follows:
    - From the dose 1 administration date for the analysis on the ES;
    - From 30 days post-dose 2 date for the analysis on the mES.
  - The end date of the follow-up time (stop) will be computed as follows:
    - Date of the last visit/contact for subjects who did not have an event;
    - Last contact date for subjects dropped out of the study, if not preceded by an event:

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

- Date of the event
- Date of HZ and/or VZV vaccination outside the study, if not preceded by an event
- The follow-up time at risk is computed using the following formula:
  - stop start + 1.

The **time at risk** will be expressed in Person-Year and derived from the follow up time (follow up time in days/365.25).



## 9.2.3. Safety

- For the analysis of HZ related complications/unsolicited AEs/SAEs/pIMDs/ concomitant medication, all vaccinated subjects will be considered and subjects who did not report an event will be considered as subjects without an event.
- AEs that need to be reported as pIMDs are listed in Table 23 of the protocol. The table presenting pIMDs, will also include the AEs considered as pIMDs as per MedDRA dictionary.
- Assessment of intensity for solicited local and general AEs will be done separately as per GSK scale and Chinese scale. From an analysis perspective, the intensity of nausea, vomiting and diarrhoea will be presented separately as per the guidelines of Chinese authorities. In addition, as per GSK standard grading, the solicited general AEs of nausea, vomiting, diarrhoea and/or abdominal pain will be presented collectively as "gastrointestinal symptoms".

For analysis as per GSK standard grading, the maximum intensity of any one of these solicited general AEs (i.e. nausea, vomiting and diarrhoea *and abdominal pain*) reported by a subject will be attributed as maximum intensity of "gastrointestinal symptoms" for that subject. Maximum of grade 3 and 4 will be considered as grade 3 *for all applicable solicited symptoms (not only gastrointestinal symptoms) in GSK standard grading table.* 

The intensity of the following solicited AEs will be assessed as described below:

Table 3 Intensity scales for solicited symptoms in adults

| Adults | | |
|---|---|---|
| Adverse Event Intensity grade | | Parameter |
| Pain at injection site | 0 | None |
| | 1 | Mild: Do not influence or do slightly influence limb activities. |
| | 2 | Moderate Influence limb activities. |
| | 3 | Severe: Influence daily life. |
| | 4 | Lose the basic selfcare ability, or hospitalization |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Temperature* | | Record temperature in °C (with 1 decimal) |
| Headache | 0 | Normal |
| | 1 | Mild: Headache that is easily tolerated |
| | 2 | Moderate: Headache that interferes with normal activity |
| | 3 | Severe: Headache that prevents normal activity |
| | 4 | Refractory; require emergency presentation or hospitalization |
| Fatigue | 0 | Normal |
| | 1 | Mild: Fatigue that is easily tolerated |
| | 2 | Moderate: Fatigue that interferes with normal activity |
| | 3 | Severe: Fatigue that prevents normal activity |
| | 4 | Emergency presentation or hospitalization |
| Gastrointestinal | 0 | Normal |
| symptom (Diarrhea) 1 Slight or transient, 3-4 times/day, stool with abnormal properties, diarrhea persisting for not more than 1 week | | |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

| | Otatistical Analysis Flan Americment |
|---|---|
| | Adults |
| Intensity | Parameter |
| grade | |
| 2 | Moderate or persistent, 5-7 times/days, stool with abnormal properties, or |
| | diarrhea >1 week |
| 3 | >7 times/day, stool with abnormal properties, or bloody diarrhea, orthostatic |
| | hypotension, electrolyte imbalance, and requiring intravenous fluid >2 L |
| 4 | Hypotensive shock, requiring hospitalization for treatment |
| 0 | Normal |
| 1 | Transient (<24 h) or intermittent, while food intake basically normal |
| 2 | Persistent nausea, leading to decreased food intake (24-48 h) |
| 3 | Persistent nausea, leading to little food intake (>48 h) or require intravenous |
| | fluid infusion |
| 4 | Life-threatening (such as hypotensive shock) |
| 0 | Normal |
| 1 | 1-2 times/24 h and do not influence activities |
| 2 | 3-5 times/24 h or activities restricted |
| 3 | >6 times within 24 h or require intravenous fluid infusion |
| 4 | Due to hypotension, require hospitalization or nutrition by other routes |
| 0 | Normal |
| 1 | Mild: Gastrointestinal symptoms that are easily tolerated |
| 2 | Moderate: Gastrointestinal symptoms that interfere with normal activity |
| 3 | Severe: Gastrointestinal symptoms that prevent normal activity |
| 0 | None |
| 1 | Mild: Myalgia that is easily tolerated |
| 2 | Moderate: Myalgia that interferes with normal activity |
| 3 | Severe: Myalgia that prevents normal activity |
| | 2<br>3<br>4<br>0<br>1<br>1<br>2<br>3<br>4<br>0<br>1<br>1<br>2<br>3<br>4<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>3<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>3<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>3<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>3<br>0<br>0<br>1<br>1<br>2<br>3<br>0<br>0<br>1<br>1<br>2<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>1<br>1<br>2<br>3<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>0<br>1<br>1<br>2<br>2<br>3<br>0<br>0<br>0<br>0<br>1<br>0 |

<sup>\*</sup> For this study, fever is defined as temperature ≥ 37.3°C as per guidelines from the Chinese authorities for axillary measurement. The preferred location for measuring temperature in this study will be the axilla.

The maximum intensity of local injection site redness/swelling will be scored at GSK using GSK's standard grading scale (based on the US Food and Drug Administration (FDA) guidelines [FDA, 2007]) and the guidelines of grading standards for AEs set by the Chinese authorities as follows.

| Grade | GSK standard grading scale | Grading scale defined by Chinese authorities |
|---|---|---|
| 0 | < 20 mm diameter | Absent |
| 1 | ≥ 20 mm to ≤50 mm diameter | 25 mm to <50 mm |
| 2 | > 50 mm to ≤100 mm diameter | 50 mm to <100 mm |
| 3 | > 100 mm diameter | >=100 mm |
| 4 | Not defined | Abscess, exfoliative dermatitis, and dermis or deep tissue necrosis* |

<sup>\*</sup>The solicited symptom diary card doesn't allow to choose grade 4 swelling or redness. Per team agreement, the grade 4 of swelling and redness will be identified when the below Preferred Terms (from MedDRA version 25.0) are reported as unsolicited adverse events within or ongoing 7 days post each dose:

- Dermatitis exfoliative
- Necrosis

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

- Skin necrosis
- Soft tissue necrosis
- Abscess
- Abscess sterile
- Abscess limb
- Abscess soft tissue

Fever will be graded as:

| Grade | GSK standard grading scale | Grading scale defined by Chinese authorities (for axillary measurement) |
|---|---|---|
| 0 | <38.0°C | <37.3°C |
| 1 | ≥38.0°C –≤38.5°C | 37.3°C – <38°C |
| 2 | >38.5°C –≤39.0°C | 38.0°C -<38.5°C |
| 3 | >39.0°C | 38.5°C - <39.5°C |
| 4 | Not defined | ≥ 39.5°C |

The preferred location for measuring temperature in this study will be the axilla. If temperature is measured by other routes (such as oral or rectal), fever grading as per GSK scale will remain the same irrespective of route of measurement. For the grading scale as per Chinese authorities, the following conversion will be used:

- Axillary temperature = Oral temperature minus 0.2°C;
- Axillary temperature = Rectal temperature minus 0.5°C.
- Axillary temperature = Tympanic membrane temperature
- For the duration of solicited adverse event within the solicited symptom follow-up or total duration, the unknown or missing end date will not be imputed.
- The definition of HZ related complication is described in section 12.5.2 of the protocol and is presented below:-

| Post-herpetic<br>neuralgia | PHN is defined by the presence of HZ-associated severe pain persisting or appearing more than 90 days after onset of the HZ rash. |
|---|---|
| Disseminated disease | Defined as $\geq$ 6 HZ lesions clearly outside the primary dermatome as per the investigator's judgment. |
| Ophthalmic disease | Defined as HZ affecting any eye structure as per the investigator's judgment. |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

| | Statistical Arialysis Flati Americinent |
|---|---|
| Neurologic<br>disease | Defined as cranial or peripheral nerve palsies, myelitis, meningoencephalitis, stroke, etc. that is temporally associated with an episode of HZ and, in the opinion of the investigator, is caused directly by VZV infection arising from the HZ episode. |
| Visceral disease | Defined as an abnormality of one or more internal organs (e.g., hepatitis, pneumonitis, gastroenteritis, etc.) that is temporally associated with an episode of HZ and, in the opinion of the investigator, is caused directly by VZV infection arising from the HZ episode |
| HZ vasculitis | Vasculopathy or vasculitis (based on clinical, laboratory or radiologic findings) that is temporally associated with an episode of HZ and, in the opinion of the investigator, is caused directly by the VZV infection arising from the HZ episode. |
| Stroke | A diagnosis of stroke requires that criteria 1, 2 and 3 are fulfilled or criteria 1 and 4 and in the opinion of the investigator is temporally associated with an episode of HZ |
| | Criterion 1: Rapid onset of localizing neurological deficit and/or change in level of consciousness; |
| | Criterion 2: Localizing neurological deficit or change in level of consciousness that lasts greater than 24 hours; |
| | Criterion 3: No other cerebral process, peripheral lesion, or other disorder is the cause of the localizing neurological deficit or change in level of consciousness; |
| | Criterion 4: Computerized Tomography (CT) scan or Magnetic Resonance Imaging (MRI) scan evidence of an acute thrombotic or hemorrhagic lesion |

• A specific COVID-19 eCRF page is used to collect any event related to COVID-19 pandemic. Input from local regulatory, local medical affairs and sites was provided to define pandemic measures periods at each site. Start date of pandemic measure period will be considered first day of month and end date of pandemic measure period will be considered as last day of month.

| | | Ι | T =: | 1 | tical Analysis Plan Amendment 1 |
|---|---|---|---|---|---|
| | | First | Start date | End date | |
| | | subject | of | of | |
| | | first visit | pandemic | pandemic | |
| | | date at | measure | measure | Reason/s for pandemic |
| Location | Center | Center | period | period | measure period |
| | | | | | Strong recommendation of mass vaccination of |
| | | | | | Covid-19 vaccines to wide population. Isolated cases in country |
| | | | M 21 | 14 21 | lack of resources that |
| | | | Mar21 | May21 | delay the Study start |
| | | | | | Covid-19 outbreak in |
| | | | | | Shanghai<br>High business, public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | region and community |
| | | | | | Citywide static |
| | | | | | management |
| | | | | | lack of resources that lead to miss of month phone |
| | | | Mar22 | Jun22 | contact |
| | | | 1/11/122 | oun22 | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Isolated cases in country |
| | | | | | Lack of resources that |
| | | | Oct22 | Nov22 | impact data entry |
| | | | | | High business public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | country Sustained community |
| | | | | | spread in geographic area |
| | | | | | local to GSK community |
| | | | | | Public health service |
| | | | | | capacity exceeded |
| | | | | | lack of resources that |
| | 248981 | 14-May-21 | Nov22 | Jan23 | impact data entry |
| | | | | | Strong recommendation of |
| | | | | | mass vaccination of |
| | | | | | Covid-19 vaccines to wide |
| | | | | | population. |
| | | | | | Isolated cases in country |
| Charact . | 240202 | 21 7-1 21 | Ma::21 | Ma21 | lack of resources that |
| Shanghai | 248302 | 21-Jul-21 | Mar21 | May21 | delay the Study start |

| | | First<br>subject<br>first visit | Start date of pandemic | End date of pandemic | |
|---|---|---|---|---|---|
| Location | Center | date at<br>Center | measure<br>period | measure<br>period | Reason/s for pandemic<br>measure period |
| Bocunon | Cemer | Conci | period | periou | Covid-19 outbreak in Shanghai High business, public life and health impact Widespread disease in region and community Citywide static management |
| | | | Mar22 | Jun22 | Lack of resources that impact data entry |
| | | | | | Province/Partial control to prevent Covid-19 Isolated cases in country |
| | | | Oct22 | Nov22 | Lack of resources that impact data entry |
| | | | Nov22 | Jan23 | High business public life and health impact Widespread disease in country Sustained community spread in geographic area local to GSK community Public health service capacity exceeded lack of resources that impact data entry |
| | | | Mar21 | May21 | Strong recommendation of mass vaccination of Covid-19 vaccines to wide population. Isolated cases in country lack of resources that delay the Study start |
| | | | | • | Covid-19 outbreak in Shanghai High business, public life and health impact Widespread disease in region and community Citywide static management Lack of resources that |
| | 248303 | 15-Jul-21 | Mar22 | Jun22 | impact data entry |

| | 1 | T | | 1 | licai Ariaiysis Pian Amendment i |
|---|---|---|---|---|---|
| | | First | Start date | End date | |
| | | subject | of | of | |
| | | first visit | pandemic | pandemic | |
| | | date at | measure | measure | Reason/s for pandemic |
| Location | Center | Center | period | period | measure period |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Isolated cases in country |
| | | | | | Lack of resources that |
| | | | Oct22 | Nov22 | impact data entry |
| | | | 00022 | 1,0,22 | High business public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | _ |
| | | | | | Country Sustained community |
| | | | | | Sustained community |
| | | | | | spread in geographic area |
| | | | | | local to GSK community |
| | | | | | Public health service |
| | | | | | capacity exceeded |
| | | | | | lack of resources that |
| | | | Nov22 | Jan23 | impact data entry |
| | | | | | Strong recommendation of |
| | | | | | mass vaccination of |
| | | | | | Covid-19 vaccines to wide |
| | | | | | population. |
| | | | | | Isolated cases in country |
| | | | | | lack of resources that |
| | | | Mar21 | May21 | delay the Study start |
| | | | | | Covid-19 outbreak in |
| | | | | | Shanghai |
| | | | | | High business, public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | region and community |
| | | | | | Citywide static |
| | | | | | management |
| | | | | | Lack of resources that |
| | | | Mar22 | Jun22 | impact data entry |
| | | | 1VI (UI 4/4 | Jun44 | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Isolated cases in country |
| | 0.45.405 | 06.7 | 0.422 | N. 66 | Lack of resources that |
| | 247421 | 06-Jun-21 | Oct22 | Nov22 | impact data entry |

| | | First | Start date | End date | |
|---|---|---|---|---|---|
| | | subject | of | of | |
| | | first visit | pandemic | pandemic | |
| | | date at | measure | measure | Reason/s for pandemic |
| Location | Center | Center | period | period | measure period |
| | | | | | High business public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | country |
| | | | | | Sustained community |
| | | | | | spread in geographic area |
| | | | | | local to GSK community |
| | | | | | Public health service |
| | | | | | capacity exceeded |
| | | | M22 | 1 22 | lack of resources that |
| | | | Nov22 | Jan23 | impact data entry |
| | | | | | Strong recommendation of |
| | | | | | mass vaccination of |
| | | | | | Covid-19 vaccines to wide |
| | | | | | population. |
| | | | | | Isolated cases in country |
| | | | | | lack of resources that |
| | | | Mar21 | Jul21 | delay the Study start |
| | | | | | Covid19 outbreak in |
| | | | | | Nanjing city and Jiangsu |
| | | | | | province |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | 7 101 | 4 21 | Lack of resources that |
| | | | Jul21 | Aug21 | delay the study start |
| | | | | | Covid-19 outbreak in |
| | | | | | Shanghai |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Lack of resources that |
| | | | Mar22 | Jun22 | delay the data entry |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Isolated cases in country |
| | | | | | Lack of resources that |
| | | | Oct22 | Nov22 | delay the data entry |
| | | | UCI22 | 110744 | |
| | | | | | High business public life |
| | | | | | and health impact |
| | | | | | Widespread disease in |
| | | | | | country |
| | | | | | Sustained community |
| Lianshui | 247564 | 11-Sep-21 | Nov22 | Jan23 | spread in geographic area |

| | | I | Ι ~ | | tical Analysis Plan Amendment 1 |
|---|---|---|---|---|---|
| | | First | Start date | End date | |
| | | subject | of | of | |
| | | first visit | pandemic | pandemic | |
| | | date at | measure | measure | Reason/s for pandemic |
| Location | Center | Center | period | period | measure period |
| Locuiton | Center | Center | periou | periou | local to GSK community |
| | | | | | Public health service |
| | | | | | capacity exceeded |
| | | | | | lack of resources that |
| | | | | | impact data entry |
| | | | | | Strong recommendation of |
| | | | | | mass vaccination of |
| | | | | | Covid-19 vaccines to wide |
| | | | | | population. |
| | | | | | Isolated cases in country |
| | | | | | lack of resources that |
| | | | Mar21 | Jul21 | delay the Study start |
| | | | | | Covid19 outbreak in |
| | | | | | Nanjing city and Jiangsu |
| | | | | | province |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Lack of resources that |
| | | | Jul21 | Aug21 | delay the study start |
| | | | 31121 | 214521 | Covid-19 outbreak in |
| | | | | | Shanghai Duaning a (Pantial a autual to |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Lack of resources that |
| | | | Mar22 | Jun22 | impact the data entry |
| | | | | | Covid-19 epidemic in |
| | | | | | Ganyu |
| | | | | | citywide static |
| | | | | | management |
| | | | | | Partial control and travel |
| | | | | | restrictions to prevent and |
| | | | | | control Covid-19 |
| | | | 1122 | 4 | lack of resources that |
| | | | Jul22 | Aug22 | impact the data entry |
| | | | | | Province/Partial control to |
| | | | | | prevent Covid-19 |
| | | | | | Isolated cases in country |
| | | | | | Lack of resources that |
| Ganyu | 248595 | 15-Sep-21 | Oct22 | Nov22 | impact the data entry |

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

| | | First<br>subject<br>first visit<br>date at | Start date of pandemic measure | End date<br>of<br>pandemic<br>measure | Reason/s for pandemic |
|---|---|---|---|---|---|
| Location | Center | Center | period | period | measure period |
| | | | | | High business public life and health impact Widespread disease in country Sustained community spread in geographic area local to GSK community Public health service capacity exceeded lack of resources that |
| | | | Nov22 | Jan23 | impact data entry |

## 10. ANNEXES

## 10.1. Business rules for standard data derivations and statistical methods

This section contains standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after study dose. If 'after study dose' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before study dose' is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

The following exceptions apply:

- Adverse event start dates with missing day: If the event starts in the same month as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after study dose) will be used to complete the date. If 'after study dose' is selected, the imputed start date will match the first (or only) study dose given during that month. If 'before study dose' is selected, the imputed date will be one day before the first (or only) study dose given during that month.
- Adverse event start dates with missing day and month: If the event starts in the same year as at least one of the study doses, the contents of AE.AESTRTPT (the flag indicating if the event occurred before or after vaccination) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first (or only) study dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first (or only) study dose given during that year.
- All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

## 10.1.2.3. Daily recording of solicited adverse events

#### 10.1.2.3.1. Studies with electronic diaries

Not applicable for the study

## 10.1.2.3.2. Studies with paper diaries

For studies using paper diaries which have questions in the CRF indicating the presence or absence of solicited events, the following rules are applicable.

- Denominators for the summary of administration site (or systemic) solicited events will be calculated using the number of participants who respond "Yes" or "No" to at least one occurrence of the specific administration site (or systemic) solicited event. If there are at least 1 non-missing value of temperature from day 1 to day 7 post vaccination, that occurrence will be counted as well in the denominator of systemic solicited events.
- When a specific solicited event is marked as having not occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=N for the specified post-dose period for the event in question), all daily measurements will be imputed as Grade 0.

212884 (ZOSTER-076) Statistical Analysis Plan Amendment 1

- For fever, if there are missing values and/or non-missing values of temperature from day 1 to day 7 post vaccination which are not qualifying fever definition per protocol for GSK intensity and Chinese intensity tables, then that subject would not be considered for 'Any' rows of the solicited event summary tables.
- When a specific solicited event is marked as having occurred following a specific study dose (i.e. SDTM CE.CEOCCUR=Y for the specified post-dose period for the event in question), any missing daily recordings will be given imputed values to allow them to contribute to the 'Any' rows but not to specific grade rows of the solicited event summary tables.
- The following table shows how participants contribute to each category for a specific solicited adverse event over the Day X to Day Y post-dose period:

| Solicited adverse event category | Participants included in the calculation of the numerator |
|---|---|
| Any | All participants with at least one occurrence of the adverse event at grade 1, 2, or 3 for table by GSK intensity scale and at grade 1, 2, 3 or 4 for table by Chinese intensity scale between Day X and Day Y or with the adverse event marked as present and at least one missing daily recording between Day X and Day Y |
| Grade 1 | All participants with at least one occurrence of the adverse event at grade 1 between Day X and Day Y |
| Grade 2 | All participants with at least one occurrence of the adverse event at grade 2 between Day X and Day Y |
| At least grade 3 | All participants with at least grade 3 or grade 4 |
| Grade 4* | All participants with at least one occurrence of the adverse event at grade 4 between Day X and Day Y |

<sup>\*</sup>this is specific to the study as grade 4 has also been defined for some solicited adverse event collected in the study as per Chinese regulation.

#### 10.1.2.4. Unsolicited adverse events

Unsolicited adverse event summaries are including serious adverse events unless specified otherwise.

Missing relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' when displayed in a statistical output.

Missing severity will follow the next imputation rules:

- If serious adverse event = 'Y' then severity = 'Severe'
- If serious adverse event = 'N' and action taken with study vaccine(s) as a result of the event = 'Dose not changed' and subject did not withdraw from the study due to this event, then severity = 'Mild'
- If previous two rules were not applicable, then severity = 'Moderate'

#### 10.1.3. Data derivation

## 10.1.3.1. Age at first dose in years

When age at first dose is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of first dose. For example:

DOB = 10SEP1983, Date of first dose = 09SEP2018 -> Age = 34 years DOB = 10SEP1983, Date of first dose = 10SEP2018 -> Age = 35 years

## 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

## 10.1.3.3. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study dose and the start date of the event. This is 1 for an event occurring on the same day as a study dose (and reported as starting after first dose).

#### 10.1.3.4. Duration of events

The duration of an event with a start and end date will be the difference between the start and end date plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the adverse event reported at grade 1 or higher during the solicited event period.

If symptom is ongoing and the end date of event is partially or fully missing, end date will not be imputed for the calculation of duration.

## 10.1.3.5. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered systemic events since the administration site flag is not included in the expedited adverse event CRF pages. Unsolicited adverse events with missing administration site flag will also be considered systemic.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

212884 (ZOSTER-076)

Statistical Analysis Plan Amendment 1

## 10.1.3.6. Counting rules for occurrences of solicited events

When the occurrences of solicited events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs.

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal except for 100% in which case no decimal will be displayed.

## 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The maximum and minimum of transformed body temperatures will be displayed with one decimal.

## 10.1.5. Statistical methodology

## 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

#### 10.2. TFL TOC

The Table Figure Listing (TFL) Table Of Content (TOC) which itemizes the planned list of TFL for final analysis with their associated lay-out is developed as a separate document.

#### 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

FDA, U.S. Department of Health and Human Services, Center for Biologics Evaluation and Research. Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. Version of September 2007.